CLINICAL TRIAL: NCT07350850
Title: In Treatment-Naive Patients With Primary Central Nervous System Lymphoma (PCNSL): A Multicenter Two-Cohort Study of Methotrexate Combined With Rituximab, Sintilimab and Pirtobrutinib (Prospective Interventional Cohort) vs. Real-World Investigator-Selected Treatment (Observational Cohort)
Brief Title: A Multicenter Two-Cohort Study of Methotrexate, Rituximab, Sintilimab and Pirtobrutinib for Treatment-Naive PCNSL vs. Real-World Investigator-Selected Treatment (Observational Cohort)
Acronym: PRIME-PCNSL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government); First Affiliated Hospital of Fujian Medical University (Other); The General Hospital of Western Theater Command (Other); China-Japan Union Hospital, Jilin University (Other)
Responsible Party: Principal Investigator, Jia Wei, chief physician, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB202512084
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PCNSL; Primary Central Nervous System Lymphoma
Keywords: Primary Central Nervous System Lymphoma (PCNSL); Methotrexate; Rituximab; Sintilimab; Pirtobrutinib; Real-World Evidence
MeSH Terms: interventions — pirtobrutinib; sintilimab; Rituximab; Methotrexate; Standard of Care

STUDY DESIGN:
Intervention Model Description: Cohort 1 (Prospective Interventional): A single-arm cohort utilizing Simon's two-stage minimax design to evaluate the efficacy and safety of the Methotrexate, Rituximab, Sintilimab and Pirtobrutinib combination. Cohort 2 (Real-World Observational): A cohort collecting real-world data (both retrospective from Sept 2023-Nov 2025 and concurrent prospective) on patients receiving investigator-selected standard-of-care (e.g., MATRix, RMT, MR-BTKi) or palliative treatments.
Who Masked: Outcomes Assessor
Masking Description: While the participants and clinical investigators are aware of the treatment assignment (Open Label), Independent radiologists (from the central imaging group) will be completely blinded to patient grouping, clinical judgment, and laboratory results when evaluating the primary endpoint (Complete Remission).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Cohort (Experimental): Patients receive Rituximab, Methotrexate, Sintilimab, and Pirtobrutinib for 6 cycles (21 days/cycle).
  Interventions: Drug: Pirtobrutinib, Sintilimab, Rituximab, Methotrexate
- Real-World Observational Cohort (Active Comparator): Participants in this cohort will receive investigator-selected standard-of-care treatments according to routine real-world clinical practice, without protocol-mandated intervention assignment. This includes: (1) Standard Treatment Subgroup: Regimens such as MATRix, RMT, or MR-BTKi. (2) Palliative Care Subgroup: Radiotherapy, low-dose chemotherapy, or supportive care.
  Interventions: Drug: Standard of Care (Investigator Selected)

INTERVENTIONS:
Drug: Pirtobrutinib, Sintilimab, Rituximab, Methotrexate — Participants in this single-arm prospective cohort will receive the investigational combination therapy: Rituximab (375 mg/m^2, IV, Day 0), Methotrexate (3.5 g/m^2, IV, Day 1; adjusted to 1.0 g/m^2 for elderly/frail patients), Sintilimab (200 mg, IV, Day 1), Pirtobrutinib (200 mg, PO, Days 1-21). Treatment cycles repeat every 21 days for up to 6 cycles.
  Arms: Interventional Cohort
Drug: Standard of Care (Investigator Selected) — Participants in the Real-World Observational Cohort receive investigator-selected treatments based on clinical guidelines. 1.Specific regimens include:
  1. MATRix: Methotrexate (3.5g/m², d1), Cytarabine (2g/m², d2-3), Rituximab (375mg/m², d0), and Thiotepa (30mg/m², d4) every 21 days .
  2. RMT: Methotrexate (3.5g/m², d1), Rituximab (375mg/m², d0), and Temozolomide (150mg/m², d1-5) every 21 days .
  3. MR-BTKi: Methotrexate (3.5g/m², d1), Rituximab (375mg/m², d0), and a covalent BTK inhibitor (Ibrutinib 560mg qd, Zanubrutinib 160mg bid, or Orelabrutinib 150mg qd) .
     2.Palliative Care Subgroup: Radiotherapy, low-dose chemotherapy, or supportive care .Radiotherapy: Low-dose Whole Brain Radiotherapy (WBRT ≤ 30Gy). Low-dose Chemotherapy: Reduced-dose Methotrexate (e.g., 1.0g/m²) or other single-agent chemotherapy. Best Supportive Care: Management of symptoms and complications without intensive anti-tumor agents.
  Arms: Real-World Observational Cohort

SUMMARY:
The goal of this clinical trial is to evaluate a new combination therapy for patients with newly diagnosed Primary Central Nervous System Lymphoma (PCNSL). The main questions it aims to answer are: (1) Does the combination of Methotrexate, Rituximab, Sintilimab, and Pirtobrutinib improve the Complete Remission Rate (CRR)? (2) Is this regimen safe and tolerable for patients? Researchers will compare this interventional group to a real-world observational group (receiving standard investigator-selected treatments) to see if the new combination improves treatment response and survival.

DETAILED DESCRIPTION:
Primary Central Nervous System Lymphoma (PCNSL) is a rare extranodal non-Hodgkin lymphoma with poor prognosis, characterized by MYD88 L265P/CD79B mutations and PD-L1/PD-L2 overexpression. Current first-line therapies based on high-dose methotrexate (HD-MTX) have limitations including high recurrence rates, poor blood-brain barrier penetration, and significant toxicity. Pirtobrutinib, a highly selective reversible BTK inhibitor, exhibits superior CNS penetration and safety profiles compared to covalent BTK inhibitors. Sintilimab (anti-PD-1) enhances anti-tumor immunity by blocking PD-1/PD-L1 axis. This study evaluates the efficacy and safety of the quadruple combination (methotrexate+rituximab + sintilimab + pirtobrutinib ) in treatment-naive PCNSL, with a real-world cohort providing comparative evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Voluntarily signed informed consent.
3. ECOG Performance Status 0-3.
4. Expected survival > 3 months.
5. Histopathologically confirmed Diffuse Large B-Cell Lymphoma (DLBCL) restricted to the CNS or eyes (PCNSL).
6. Measurable lesion on contrast-enhanced MRI (>10x10 mm) or positive CSF cytology for leptomeningeal disease.
7. No prior systemic treatment for lymphoma (corticosteroids excepted).
8. Adequate bone marrow and organ function (ANC >=1.5x10^9/L, PLT >=80x10^9/L, Hb >=80 g/L; Bilirubin <=1.5xULN, AST/ALT <=2.5xULN; Creatinine <=1.5xULN or CrCl >=60 mL/min) .
9. Stable controlled comorbidities allowed (e.g., hypertension with blood pressure <=160/100 mmHg, type 2 diabetes with HbA1c <=8%, mild coronary heart disease without myocardial infarction in the past 6 months).
10. Basic communication ability to complete PROs questionnaires (no severe cognitive impairment).
11. Reproductive-aged females and males with childbearing potential: No pregnancy plans during the study and 3 months after treatment discontinuation; use effective contraception (abstinence, physical contraception, or hormonal contraceptives initiated >=3 months before first dose). Males prohibited from donating sperm during treatment and 3 months after discontinuation.
12. For Observational Cohort (Palliative Care Subgroup only): Pathologically confirmed DLBCL restricted to the CNS or eyes; Follow-up available for efficacy assessment (at least one CR evaluation) .

Exclusion Criteria:

1.Prior treatment with PD-1/PD-L1 inhibitors or CTLA4 monoclonal antibodies. Uncontrolled active infection. 2.Uncontrolled or significant cardiovascular diseases: 3.Congestive heart failure (NYHA class III/IV),

1. myocardial infarction, unstable angina within 6 months before first dose; arrhythmia requiring treatment; LVEF <50%.
2. Primary cardiomyopathy.
3. History of clinically significant QTc prolongation, second-degree type II/third-degree atrioventricular block, or QTc interval (Fridericia method) >470 msec (females) / >480 msec (males).
4. Atrial fibrillation (EHRA grade ≥2b).
5. Refractory hypertension. 4.Active hepatitis B/C infection (HBV-DNA ≥ detection limit, HCV RNA positive) or syphilis. (Exceptions: HBV-DNA < detection limit, cured HCV).

5.HIV infection. 6.Prior organ transplantation or allogeneic stem cell transplantation. 7.Pregnant or lactating females. 8.Prior/current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, or radiation pneumonitis (unsuitable for study per investigator).

9.Autoimmune diseases requiring systemic treatment within 2 years. 10.For Observational Cohort (Palliative Care Subgroup only): Incomplete clinical data (e.g., no pathological report, inability to perform MRI/PET-CT assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | At the completion of induction treatment(approximately 18 weeks)
  Proportion of participants achieving Complete Response (CR) at the end of treatment. Efficacy is evaluated by both investigators and independent imaging personnel based on the International Primary CNS Lymphoma Collaborative Group (IPCG) criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At the completion of induction treatment (approximately 18 weeks)
  Sum of Complete Response (CR) and Partial Response (PR) rates.
Duration of Response (DOR) | Up to 2 years.
  Time from documentation of tumor response (CR or PR) to disease progression or death.
Disease Control Rate (DCR) | At the completion of induction treatment (approximately 18 weeks)
  The proportion of patients whose tumor is controlled (no progression or shrinkage), defined as the sum of Complete Response (CR), Partial Response (PR), and Stable Disease (SD) rates.
Progression-Free Survival (PFS) | Up to 2 years.
  The time interval from the start of treatment to tumor progression (PD) or death from any cause.
Overall Survival (OS) | Up to 5 years as per long-term follow-up mentions
  The time from confirmed diagnosis to death from any cause.
Overall Survival Rate (OS Rate) | 1 year.
  The percentage of surviving patients out of the total number of included patients (specifically assessed as 1-year OS rate in study objectives).
Safety and Tolerability (Adverse Events) | Throughout the study process, up to 30 days after the last dose.
  Assessment of safety based on the severity grading of Adverse Events (AE) according to NCI CTCAE v5.0. This includes evaluation via physical examination, vital signs, performance status, ECG, laboratory tests, and AE severity.
Patient Reported Outcomes (PRO) | Baseline, every 2 cycles (approximately week 6 and week 12) during treatment, at treatment completion (approximately week 18), and every 3 months during follow-up for up to 2 years
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The questionnaire consists of 30 items, with scores ranging from 0 to 100. For functional scales (e.g., physical, role functioning) and the global health status, a higher score represents a better level of functioning or quality of life. For symptom scales/items (e.g., fatigue, nausea), a higher score represents a worse outcome or greater symptom burden

OTHER OUTCOMES:
Correlation between Molecular Subtypes and Treatment Response (CRR) | Through study completion, an average of 1 year.
  To evaluate the correlation between molecular subtypes (defined by MYD88 L265P and CD79B mutation status) and the Complete Response Rate (CRR). Mutation status is assessed via Next-Generation Sequencing (NGS). Treatment response is assessed by investigators and independent radiologists using the International Primary CNS Lymphoma Collaborative Group (IPCG) criteria based on brain MRI .

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No